CLINICAL TRIAL: NCT05525663
Title: Physical Rehabilitation for Older Patients With Acute Heart Failure With Preserved Ejection
Brief Title: Physical Rehabilitation for Older Patients With Acute Heart Failure With Preserved Ejection Fraction
Acronym: REHAB-HFpEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00087718; R01AG078153 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation Intervention (Experimental): The Rehabilitation Intervention is a novel, progressive, multi-domain rehabilitation and exercise training intervention. The intervention will include strength, balance, endurance, and mobility training and the specific training exercises will be tailored based on participant performance in each of these domains. The intervention will begin as soon as possible after randomization during the hospitalization and will continue 3 times per week in an outpatient setting for 12 weeks.
  Interventions: Behavioral: Rehabilitation Intervention
- Attention Control (No Intervention): Attention control participants are contacted bi-weekly by study staff to maintain contact, collect information regarding health status, clinical events, and physical activity/exercise, and ensure retention; they do not receive any specific exercise recommendations.

INTERVENTIONS:
Behavioral: Rehabilitation Intervention — progressive, multi-domain rehabilitation and exercise training intervention
  Arms: Rehabilitation Intervention

SUMMARY:
The REHAB-HFpEF trial will determine whether a novel physical rehabilitation intervention will improve the primary outcome of combined all-cause rehospitalizations and mortality and the secondary outcome of major mobility disability during 6-month follow-up in patients hospitalized for heart failure and preserved ejection fraction (HFpEF), which is nearly unique to older persons, and for which there are few treatment options.

DETAILED DESCRIPTION:
REHAB-HFpEF, is a multicenter, randomized, attention-controlled, single-blind trial to examine the hypothesis that, a novel, tailored, progressive, multi-domain physical rehabilitation intervention administered to older patients with acute decompensated heart failure (ADHF) with preserved ejection fraction (HFpEF) beginning early during hospitalization and continuing for 12 weeks in a structured outpatient setting, and continuing as a maintenance program will reduce the rate of combined all-cause rehospitalization and death at 6 months (the primary outcome), and reduce major mobility disability (MMD) prevalence at 6 months (the secondary outcome). This trial, REHAB-HFpEF, builds upon preliminary studies, including the phase 2 REHAB-HF trial, which suggests this intervention may yield significant benefits for this population which are largely older, frail, and with few evidence-based treatment options. Participants will be recruited from 20 clinical centers, each of which may have up to 3 tightly-affiliated 'satellite' sites geographically-close, under their direct management. Together, these centers will recruit a total of 880 consenting patients >=60 years old hospitalized with ADHF with HFpEF. Following informed consent and baseline testing, the participants will be randomized in a 1:1 fashion to receive a novel, progressive, multi-domain rehabilitation and exercise training intervention or attention control. The intervention will include strength, balance, endurance, and mobility training and the specific training exercises will be tailored based on participant performance in each of these domains. The intervention will begin as soon as possible after randomization during the hospitalization and will continue 3 times per week in an outpatient setting for 12 weeks. Those randomized to the attention control will be contacted bi-weekly by study staff to maintain contact, collect information regarding health status, clinical events, and physical activity/exercise, and ensure retention; they do not receive any specific exercise recommendations. Both arms will receive all services ordered by their primary physician (usual care) and undergo measures of physical function, cognitive function, and quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

1. Age >=60 years old
2. Ejection Fraction >=45%
3. In the hospital setting >24 hours for the management of acute decompensated heart failure (ADHF), or diagnosed with ADHF after being hospitalized for another reason. ADHF will be confirmed by the site physician, and will be defined according to the Food and Drug Administration (FDA) definition of hospitalized heart failure as a combination of symptoms, signs, and HF-specific medical treatments, and requires that all 4 of the following are met:

   * At least 1 symptom of HF which has worsened from baseline: a. dyspnea at rest or with exertion; b. exertional fatigue; c. orthopnea; d. paroxysmal nocturnal dyspnea (PND)
   * At least 2 of the following signs of HF: a. Pulmonary congestion or edema on physical exam (rales or crackles) or by chest X-ray; b. Elevated jugular venous pressure or central venous pressure >=10 mm Hg; c. peripheral edema; d. wedge or left ventricular end diastolic pressure >=15 mmHg; e. rapid weight gain (>=5 lbs.); f. Increased b-type natriuretic peptide (BNP) (>=100 pg/ml) or N-terminal prohormone BNP (>=220pg/ml)
   * Change in medical treatment specifically targeting HF, defined as change in dose or initiation of or augmentation of at least 1 of the following therapies: a. diuretics; b. vasodilators; c. other neurohormonal modulating agents, including angiotensinconverting enzyme inhibitors, angiotensin II receptor blockers (with or without neprilysin inhibitor), beta-blockers, aldosterone inhibitors, direct renin inhibitors, or sodium-glucose co-transporter-2 inhibitors
   * The primary cause of symptoms and signs is judged by the investigator to be due to HF
4. Adequate clinical stability to allow participation in study assessments and the intervention Independent with basic activities of daily living, including the ability to ambulate independently (with or without the use of an assistive device) prior to admission
5. Able to walk 4 meters (with or without the use of an assistive device) at the time of enrollment

Exclusion Criteria:

1. Acute myocardial infarction within the past 3 months, or planned coronary artery intervention (percutaneous or surgical) within the next 6 months (Note: given that cardiac biomarkers such as troponin are frequently elevated in HF patients, the diagnosis of acute myocardial infarction should be based on clinical diagnosis, not biomarkers alone)
2. Severe aortic or mitral valve stenosis
3. Severe valvular heart disease with planned intervention within next 6 months
4. Known pericardial constriction, genetic hypertrophic cardiomyopathy, or infiltrative cardiomyopathy including amyloid heart disease (amyloidosis)
5. Planned discharge other than to home or a facility where the participant will live independently
6. Terminal illness other than HF with life expectancy <1 year
7. Impairment from stroke or other medical disorders that preclude participation in the intervention
8. Known dementia by medical record documentation, OR patients with Montreal Cognitive Assessment (MoCA) <=18 AND without social support, OR MoCA <10 regardless of social support
9. Advanced chronic kidney disease defined as estimated glomerular filtration rate <20 mL/min/1.73 m2 or on chronic or intermittent dialysis or dialysis anticipated within the next 6 months
10. Already engaging in regular moderate to vigorous exercise conditioning defined as >30 minutes per day, >= twice per week consistently during the previous 6 weeks
11. Enrollment in a clinical trial not approved for co-enrollment
12. High risk for non-adherence as determined by screening evaluation
13. Inability or unwillingness to comply with the study requirements or give consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Combined All-cause Rehospitalization and Death | Month 6
  Rate of combined all-cause rehospitalizations and death 6 months following discharge from index hospitalization.

SECONDARY OUTCOMES:
Prevalence of major mobility disability (MMD) | Month 6
  Percentage of participants with MMD, defined as the inability to walk 160 meters during a 6 minute walk test.

OTHER OUTCOMES:
All-cause rehospitalization | Month 6
  Exploratory outcome. Rate of rehospitalizations 6 months following discharge from index hospitalization.
All-cause death | Month 6
  Exploratory outcome. Rate of death 6 months following discharge from index hospitalization.
Cardiovascular rehospitalization and death | Month 6
  Exploratory outcome. Rate of combined cardiovascular rehospitalizations and death 6 months following discharge from index hospitalization.
Short Physical Performance Battery (SPPB) | Month 6
  Exploratory outcome. The Short Physical Performance Battery is scored on a scale of 0-12, with a higher score indicating better physical function.
6-minute Walk Distance (6MWD) | Month 6
  Exploratory outcome. Distance walked in 6 minutes.
Quality of Life Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) | Month 6
  Exploratory outcome. The KCCQ is a heart failure disease-specific quality of life measure encompassing domains of physical limitation, HF symptoms, quality of life, and social limitation scored on a scale of 0-100 with higher scores indicating better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W Kitzman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No